CLINICAL TRIAL: NCT05837208
Title: Determination of the Thickness Truly Applied of the SPRAY50+ on Different Areas of the Face Estimated by a Multispectral Imaging Method, After Application of the Product With and Without Recommendations of Use by a Group of Healthy Subjects
Brief Title: Determination of Product Thickness Applied on Different Areas of the Face Using a Multispectral Imaging Method
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: ADPROTECTPF
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Sunscreen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated Group: all subjects will apply the study product RV4369A
  Interventions: Other: RV4369A cosmetic product

INTERVENTIONS:
Other: RV4369A cosmetic product — The product is applied 1 or 2 times during the 2 study visits. The product is recovered by the technician after application of the product by the volunteer.
  Application modalities:
  Inclusion Assessment: The study product is given to the volunteer who applies it to his face (forehead) according to his usual habits.
  After a waiting time and Multispectral camera measurements, the study product is again applied by the volunteer to his face according to his usual habits.
  Final assessment: The study product is applied by the Clinical Research Technician on the subject's forearm on 4 delimited areas at specific quantities.
  After a waiting period and Multispectral camera measurements on the forearm areas, the study product is given to the volunteer who applies it on his face according to the recommendations of use provided by the Technician.

SUMMARY:
The aim of the study is to determine:

* the thickness of the RV4369A truly applied on different areas of the face after single application of the product determined by a multispectral imaging method.
* the influence of a second application of the product 15 to 30 minutes after the first application on the product thickness determined by multispectral imaging method.
* the influence of the recommendations of use provided to the subjects before application of the product on the product thickness determined by multispectral imaging method .

DETAILED DESCRIPTION:
This study is a monocentric, comparative, open study performed on the face and forearms of healthy adults.

Planning of the visits:

Visit 1: Inclusion visit (D1) Visit 2: End of study visit (D10), a window of +/- 2 days is allowed for this evaluation, * The theoretical study duration for each subject is 10 days. The maximal study duration for each subject is 12 days.

ELIGIBILITY:
Inclusion Criteria:

* Dry, normal to combination skin
* Phototype I to V inclusive.
* Absence of significant facial hair.

Exclusion Criteria:

Population

* Pregnant, breastfeeding women.
* For men: moustached or bearded.
* Substantial hair on the forearm and face.
* Application of keratolytic or self-tanning products to the face, forearms and arms in the four weeks prior to inclusion.
* With scars or other cutaneous characteristics, sunburn on forearms in the test areas, the size of which is considered incompatible with the study.
* Application of water, cleansing or beauty products to the forearms and arms since the last wash on the evening before inclusion.

Diseases :

* Known history of allergy to any of the investigational product ingredients.
* Known history of allergy to latex.
* Skin lesions or skin disease on the face or on the arms and forearms that may affect test results (seborrheic dermatitis, atopic dermatitis, psoriasis, acne, rosacea, etc.).

Treatments:

* Ongoing local or Oral treatment (retinoids, anti-inflammatory) that may affect test results.

Ages: 20 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Panel of healthy volonteers
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Amounts of sun spray applied to the face, measured by multispectral imaging after single application by the subject | Visit 1 (Day 1)
  The product quantity applied by the subject (mg/cm2) will be extrapolated from a reference curve build using an image analysis technique
Amounts of sun spray applied to the face, measured by multispectral imaging after 2 applications by the subject | Visit 1 (Day 1)
  The product quantity applied by the subject (mg/cm2) will be extrapolated from a reference curve build using an image analysis technique
Amounts of sun spray applied to the face, measured by multispectral imaging after 1 application by the subject and according to the recommendations of use provided by the technician | Visit 2 (Day 10)
  The product quantity applied by the subject (mg/cm2) will be extrapolated from a reference curve build using an image analysis technique
Comparisons between measurements of sun spray amounts determined by multispectral imaging | Visit 1 (Day1) and visit 2 (Day 10)
  Comparaisons between an application without recommendations of use (Visit 1), an application without recommendations followed by a second application (Visit 1) and an application according to the recommendations of use (Visit 2)

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse Nocera, MD, Principal Investigator — Pierre Fabre Dermo Cosmetique
Locations (1):
- Skin Research Center, Toulouse, France